CLINICAL TRIAL: NCT04272853
Title: Sex and Sleep: Perception of Sex as a Possible Factor for Sleep Promotion in a Population of Athletes
Brief Title: Sex & Sleep in Athletes
Acronym: Sex&Sleep
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: Sex&Sleep
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2020-02

CONDITIONS: Sexual Behavior; Sleep; Sport Injury
Keywords: Athlete; Exercise; Training Load
MeSH Terms: conditions — Sexual Behavior; Motor Activity | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Athletes: 164 subjects will be recruited (see calculation of the sample size for details): all subjects will be athletes, professional or non-professional, belonging to any sporting discipline, members of one of the sports federations of the Lombardy region, officially recognized by CONI (National Committee of Italian Olympic Team).
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Compilation of the interview concerning: demographic data, sports practice, habits on sleep, sexual habits, perception of the relationship between sexual habits and sleep, perception of the relationship between sexual habits and sports practice.

SUMMARY:
Achieving the correct quantity and quality of sleep is essential for the health and recovery processes of the athlete; night rest is often negatively influenced by many variables, including: high training loads, long-range trips, evening competitions, and / or high levels of anxiety and stress. High training loads can therefore have negative influences both on sleep but also on the risk of injury in athletes. Understanding and studying, in different sports, how sexual / masturbatory activity can influence sleep has primary importance for athletic and medical staff of athletes with the ultimate aim of preserving sports performance and reducing the risk of injuries. The primary objective of this experimentation is to explore the perceived relationship between sexual activity (or masturbation), sleep quality and sleep latency in a population of athletes.

DETAILED DESCRIPTION:
Achieving the correct quantity and quality of sleep is essential for the health and recovery processes of the athlete; night rest is often negatively influenced by many variables, including: high training loads, long-range trips, evening competitions, and / or high levels of anxiety and stress. High training loads can therefore have negative influences both on sleep but also on the risk of injury in athletes. Understanding and studying, in different sports, how sexual / masturbatory activity can influence sleep has primary importance for athletic and medical staff of athletes with the ultimate aim of preserving sports performance and reducing the risk of injuries.

The primary objective of this experimentation is to explore the perceived relationship between sexual activity (or masturbation), sleep quality and sleep latency in a population of athletes. To achieve this goal, the subjects will compile an interview, concerning: demographic data, sports practice, sleep habits, sexual habits, perception of the relationship between sexual habits and sleep, perception of the relationship between sexual habits and sport. In addition, data will be collected regarding honesty and embarrassment in completing the interview.

Secondary study aims are:

1. Evaluate the possible differences in the perceived relationship between sexual activity and sleep quality / latency in relation to the gender of the athletes.
2. Evaluate the possible differences in the perceived relationship between sexual activity and sleep quality / latency in different sports disciplines.
3. Evaluate the differences in the perceived relationship between sexual activity and sleep quality / latency in professional and non-professional athletes.
4. Evaluate the differences in habits concerning night rest between individual and team sports athletes.
5. Evaluate the honesty and embarrassment rate when completing the interview.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female sex, of any ethnicity;
2. Age between 18 and 40;
3. Cognitively intact;
4. Amateur or professional athletes;
5. Practicing any type of sport for at least 6 years, for at least 4 hours a week.
6. Members with one of the sports federations of Lombardy, officially recognized by CONI.
7. Signature and acceptance of informed consent to collaborate in all the procedures necessary for the study.

Exclusion Criteria:

1. Subjects under 18;
2. Shift or part-time worker;
3. Use of drugs and / or supplements able to influence sleep (eg: melatonin);
4. Any clinical condition (eg: musculoskeletal injury), diagnosed by a sports doctor or orthopedist, which does not guarantee the athlete to train;
5. Active smoke;
6. Non-acceptance of informed consent.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is represented by the athletes, professional and non-professional, of the Lombardy region and members of one of the sports federations officially recognized by CONI.
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Perception of the relationship between sexual habits and sleep | hrough study completion, an average of 1 year
  The perception is assessed by the interview and is expressed in "improved" or "equal to" or "decreased" compared to normal sleep routines

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No